CLINICAL TRIAL: NCT03114735
Title: The Effects of Preoperative Anxiety and Pain Sensitivity on the Intraoperative Hemodynamics, Consumption of Propofol and Postoperative Recovery in Cases of Endoscopic Ultrasonography (EUS) Received Sedoanalgesia
Brief Title: Effects of Preoperative Anxiety and Pain Sensitivity in Cases of Endoscopic Ultrasonography Received Sedoanalgesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ferda Yilmaz Inal, Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 71306642-050.01.04-21/28
Record Dates: First submitted 2017-03-25; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Sedoanalgesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The objective of this study was to detect whether preoperative anxiety and pain sensitivity had effects on the consumption of anesthetics, time to achieve desired level of sedation, patient and endoscopist satisfaction, and postoperative recovery time and pain in deep sedation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 category
* between the ages of 20 and 65
* patients who has an education level and mental state to complete the scale and questionnaire provided for assessment

Exclusion Criteria:

* patients who has a psychiatric and neurological disease and use psychiatric drugs and chronic alcohol intake

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective endoscopic ultrasonography with deep sedation
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2017-05-01 (Estimated); Study Completion 2017-06-01 (Estimated)

PRIMARY OUTCOMES:
consumption of propofol(mg) | 1-3 hours
  initial dose infusion of 1 mg.kg-1 , maintenance dose 2 mg/kg/h, additional dose 0,1mg/kg in case of insufficient sedation
the heart rate(n/min) | 1-3 hours
  During procedure
arterial pressure(mmHg) | 1-3 hours
  During procedure
peripheral oxygen saturation(%) | 1-3 hours
  during procedure
postoperative nausea and vomiting (Numeric Rank Score) | 1-3 hours
  After procedure
Post-procedure pain(Visual Analog Score) | 1-3 hours
  After procedure

REFERENCES:
- [Derived] Yilmaz Inal F, Yilmaz Camgoz Y, Daskaya H, Kocoglu H. The Effect of Preoperative Anxiety and Pain Sensitivity on Preoperative Hemodynamics, Propofol Consumption, and Postoperative Recovery and Pain in Endoscopic Ultrasonography. Pain Ther. 2021 Dec;10(2):1283-1293. doi: 10.1007/s40122-021-00292-7. Epub 2021 Jul 22. PMID 34292516